CLINICAL TRIAL: NCT03315013
Title: Randomized Evaluation of a Revised, Simplified Clinical Algorithm for Identifying Patients Eligible for Immediate Initiation of Antiretroviral Therapy for HIV (SLATEII)
Brief Title: Revised Simplified Algorithm for Treatment Eligibility for HIV (SLATEII)
Acronym: SLATEII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: University of Witwatersrand, South Africa (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Sydney Rosen, Professor, BUSPH, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-37010; OPP1136158 (Other Grant/Funding Number: Bill and Melinda Gates Foundation); 4852 (Registry Identifier: NHREC South Africa); 171011 (Other: HREC (Medical) Wits University)
Record Dates: First submitted 2017-10-06; First posted 2017-10-19 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: HIV/AIDS; Antiretroviral Therapy
Keywords: Antiretroviral therapy initiation; Sub-Sahara Africa; ART
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLATE (Experimental): The SLATE arm will be administered the SLATE II algorithm and initiated on ART immediately if eligible under the algorithm. Patients not eligible under the algorithm will be referred for standard care.
  Interventions: Procedure: SLATE II
- Standard (No Intervention): The standard arm will be referred to standard care after study enrollment.

INTERVENTIONS:
Procedure: SLATE II — The SLATE II algorithm is a series of questions and procedures that allow a study clinician to determine if antiretroviral therapy for HIV can be started immediately (same-day) or if additional care or services are needed before ART initiation.
  Other Names: Revised Simplified Algorithm for Treatment Eligibility
  Arms: SLATE

SUMMARY:
In its 2017 revision of the global guidelines for HIV care and treatment, the World Health Organization called for rapid or same-day initiation of antiretroviral treatment (ART) for eligible patients testing positive for HIV. In sub-Saharan Africa, where most HIV patients are located, studies continue to document high losses of treatment-eligible patients from care before they receive their first dose of antiretroviral medications (ARVs). Among facility-level reasons for these losses are treatment initiation protocols that require multiple clinic visits and long waiting times before a patient who tests positive for HIV is dispensed an initial supply of medications. Simpler, more efficient, accelerated algorithms for ART initiation are needed, including strategies for rapid initiation in patients with symptoms of tuberculosis, most of whom do not have active TB.

In July 2017, the original SLATE study (SLATE I) completed enrollment in South Africa. One of the most striking findings of the study so far is the large proportion of patients who "screened out" of the SLATE algorithm and were referred for additional services rather than started on ART immediately. Among 298 patients assigned to the intervention arm and evaluated for immediate treatment eligibility under the SLATE algorithm, 149 (50%) screened out, two thirds of these (100/149) due to symptoms of TB. The vast majority of the TB suspects (93/100, 93%) tested negative for active TB.

The SLATE II study will revise the original SLATE algorithm to provide a pathway for immediate ART initiation for some patients with TB symptoms. Under SLATE II, patients with TB symptoms will be clinically evaluated by the study nurse and will receive a urine point of care LAM (lipoarabinomannan antigen of mycobacteria) test. Those with milder symptoms and a negative LAM test will be offered immediate ART. Those with more serious symptoms and/or a positive LAM test will be asked to return the next day to receive TB test results and either immediate ART or TB treatment. All intervention arm patients (symptomatic and asymptomatic) will be asked for a sputum sample for Xpert testing, and positives will be contacted on the next day. The SLATE II algorithm will also incorporate other improvements identified from SLATE I.

DETAILED DESCRIPTION:
SLATE II is be a pragmatic, individually randomized evaluation to determine the effectiveness of the revised algorithm in increasing ART initiation, compared to standard care, among non-pregnant adult patients. Six hundred HIV-infected adult patients not yet on ART will be enrolled during a routine clinic visit and randomized to receive the intervention or standard care. Patients in the intervention arm will be administered a revised version of the SLATE screens, including the TB add-on; those found eligible under the algorithm will be offered immediate treatment initiation, while those who are not eligible will be referred for standard clinic care. Patients in the standard arm will be referred for ART initiation under standard clinic procedures. All care after the initial visit will be by the clinic under standard care. Primary outcomes will be ART initiation within 7 days of study enrollment and viral suppression within 8 months of study enrollment.

The study is being conducted at three healthcare facilities (clinics) in South Africa. In September 2017, the South African National Department of Health instructed all clinics to offer same-day ART initiation to eligible patients but provided little guidance on determining eligibility. SLATE II will help to create such guidance. If successful, it will improve on the SLATE approach to collecting and interpreting a minimum set of patient data that will avoid delaying treatment initiation for the majority of patients who are eligible for immediate ART, while deferring initiation in the minority who should not start immediately.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) (initiating children and adolescents on ART is likely to require additional information and adherence support, making the SLATE algorithm less applicable to pediatric populations)
* Confirmed HIV-positive test result at any time (may have been diagnosed previously)
* Self-report that patient is not currently on ART and has not been prescribed ART in the past three months
* Presented at the study clinic for any HIV-related reason or other reason that led to referral for HIV testing or care

Exclusion Criteria:

* Pregnant (pregnancy is an exclusion criterion because treatment guidelines for pregnant women differ from those for non-pregnant adults; most pregnant women are diagnosed with HIV and initiated on ART in antenatal clinics, not general adult HIV clinics)
* Not intending to return to this clinic for further HIV care in the coming year (i.e. intends to seek further care somewhere else)
* Not willing to be traced by phone or in person for follow-up care if test results received after the enrollment visit indicate that further care is needed
* Not physically, mentally, or emotionally able to participate in the study, in the opinion of the investigators or study staff
* Not willing or able to provide written informed consent to participate in the study
* Previously enrolled in the same study or the SLATE I study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients initiated on ART | 7 days after study enrollment
  % of enrolled patients initiated onto ART within one week of study enrollment, which may occur at HIV diagnosis or at a pre-ART follow-up visit
Proportion of patients initiated on ART and alive, in care, and retained | 8 months after study enrollment
  Proportion of enrolled patients initiated on ART within 28 days of study enrollment and retained in care 8 months after study enrollment, as indicated by a clinic visit no more than 7 months after ART initiation

SECONDARY OUTCOMES:
Proportion of TB suspects initiated on ART within 14 days of study enrollment | 14 days after study enrollment
  Proportion of TB suspects initiated on ART within 14 days of study enrollment
Proportions of patients initiated on ART within 1, 14, and 28 days of study enrollment | 28 days after study enrollment
  Proportions of patients initiated on ART within 1, 14, and 28 days of study enrollment
Proportions of all patients and of TB suspects who initiate ART and are virally suppressed eight months after having an HIV test or enrolling in HIV care | 8 months after study enrollment
  Viral suppression stratified by TB symptom status at baseline
Proportions of all patients and of TB suspects who initiate ART and are alive, in care, and retained on ART 14 months after having an HIV test or enrolling in HIV care | 14 months after study enrollment
  Retention 12 months after enrollment, allowing 1 month for initiation and 1 month for making and recording data from 12-month visit.
Proportions of HIV-positive patients presenting at study clinics and not yet on ART who are eligible and ineligible for immediate initiation using SLATE algorithm criteria | 1 day after study enrollment
  Patients who screen in and screen out of algorithm in intervention arm
Reasons for ineligibility for immediate initiation | 1 day after study enrollment
  Reasons for ineligibility for immediate initiation, among those found ineligible in the intervention arm
Median time to ART initiation (days) for each arm | 28 days after study enrollment
  Median and IQR time to ART initiation (days) for each arm
Adverse events | 1, 7, 14, and 28 days after enrollment; 8 and 14 months after enrollment
  Frequency and types of adverse events reported in medical records after ART initiation for each follow up period
Patient preferences | 1 day after enrollment
  Patient self-reported preferences on the speed and timing of ART initiation, from questionnaires
LAM test results | 1 day after enrollment
  Proportion of symptomatic patients who test positive for TB using the LAM test
Xpert test results | 1 week after enrollment
  Proportions of symptomatic and asymptomatic patients who test positive for TB using Xpert MTB/RIF, among those able to produce a sputum sample
Costs to patients | 14 months after study enrollment (end of followup)
  Costs to patients of ART initiation under standard and intervention procedures
Costs to providers | 14 months after study enrollment (end of followup)
  Costs to providers of ART initiation under standard and intervention procedures
Differences from SLATE I | 14 months after study enrollment (end of followup)
  Comparison of results of SLATE II study to SLATE I study

CONTACTS AND LOCATIONS:
Overall Officials: Sydney B Rosen, Principal Investigator — Boston University
Locations (1):
- Health Economics and Epidemiology Research Office, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
After protocol closure, dis-identified data generated by the study will be shared on Dryad. Data from patients' medical records do not belong to the study and cannot be shared but may be available on request from the study sites.
Supporting Information: Study Protocol, ICF
Time Frame: After protocol closure, which will occur approximately one year after all study outcomes have been reached.

REFERENCES:
- [Background] Brennan AT, Maskew M, Larson BA, Tsikhutsu I, Bii M, Vezi L, Fox MP, Venter WD, Ehrenkranz P, Rosen S. Who is seeking antiretroviral treatment for HIV now? Characteristics of patients presenting in Kenya and South Africa in 2017-2018. J Int AIDS Soc. 2019 Sep;22(9):e25358. doi: 10.1002/jia2.25358. PMID 31518058
- [Background] Brennan A, Maskew M, Larson BA, Tsikhutsu I, Bii M, Vezi L, Fox M, Venter WDF, Ehrenkranz PD, Rosen S. Prevalence of TB symptoms, diagnosis and treatment among people living with HIV (PLHIV) not on ART presenting at outpatient clinics in South Africa and Kenya: baseline results from a clinical trial. BMJ Open. 2020 Sep 6;10(9):e035794. doi: 10.1136/bmjopen-2019-035794. PMID 32895266
- [Background] Scott NA, Maskew M, Fong RM, Olson IE, Brennan AT, Fox MP, Vezi L, Ehrenkranz PD, Rosen S. Patient Perspectives of Quality of the Same-Day Antiretroviral Therapy Initiation Process in Gauteng Province, South Africa: Qualitative Dominant Mixed-Methods Analysis of the SLATE II Trial. Patient. 2021 Mar;14(2):175-186. doi: 10.1007/s40271-020-00437-4. PMID 32909218
- [Background] Rosen S, Maskew M, Brennan AT, Fox MP, Vezi L, Ehrenkranz PD, Venter WDF. Improved simplified clinical algorithm for identifying patients eligible for immediate initiation of antiretroviral therapy for HIV (SLATE II): protocol for a randomized evaluation. Trials. 2018 Oct 11;19(1):548. doi: 10.1186/s13063-018-2928-5. PMID 30305142
- [Result] Maskew M, Brennan AT, Fox MP, Vezi L, Venter WDF, Ehrenkranz P, Rosen S. A clinical algorithm for same-day HIV treatment initiation in settings with high TB symptom prevalence in South Africa: The SLATE II individually randomized clinical trial. PLoS Med. 2020 Aug 27;17(8):e1003226. doi: 10.1371/journal.pmed.1003226. eCollection 2020 Aug. PMID 32853271
- [Derived] Maskew M, Parrott S, De Voux L, Sharpey-Schafer K, Crompton T, Govender AC, Pisa PT, Rosen S. Triaging Clients at Risk of Disengagement from HIV Care: Application of a Predictive Model to Clinical Trial Data in South Africa. Risk Manag Healthc Policy. 2025 May 16;18:1601-1619. doi: 10.2147/RMHP.S510666. eCollection 2025. PMID 40395656
- [Derived] Maskew M, Brennan AT, Venter WDF, Fox MP, Vezi L, Rosen S. Retention in care and viral suppression after same-day ART initiation: One-year outcomes of the SLATE I and II individually randomized clinical trials in South Africa. J Int AIDS Soc. 2021 Oct;24(10):e25825. doi: 10.1002/jia2.25825. PMID 34612601

DOCUMENTS (1):
  • Study Protocol (2017-10-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT03315013/Prot_001.pdf